CLINICAL TRIAL: NCT05737446
Title: Oxygen Partial Pressure After Breast Cancer Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 07068-02
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Surgery-Complications; Hypoxia
Keywords: Breast cancer surgery; postoperative hypoxia; Lung function
MeSH Terms: conditions — Breast Neoplasms; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypoxia and reduced oxygen partial pressure is commonly occurring after abdominal surgery. This study aims to investigate whether similar changes also occur after breast cancer surgery.

Inclusion: 60 women undergoing breast cancer surgery. Exclusion: Dementia or cognitive impairment that makes it impossible to participate in the study.

Arterial blood gas and lung function are undertaken before surgery and the day after surgery

DETAILED DESCRIPTION:
Postoperative hypoxia complicates 30% - 50% of abdominal surgeries. People at particular risk for postoperative pulmonary complications including severe hypoxia are those who undergo abdominal surgery, emergency surgery or have a respiratory failure due to chronic lung disease. The cause of postoperative hypoxia and reduced lung function is unknown. Previous studies report that arterial partial pressure (PaO2) decreased by an average of 2 kilopascal after abdominal surgery, while carbon dioxide partial pressure (PaCO2) was unchanged and vital capacity decreased by 35%. The effect of breast cancer surgery on oxygen and carbon dioxide partial pressure and lung function has to the best of the investigators knowledge not been investigated. This study aims to investigate possible changes in oxygen partial pressure, carbon-dioxide partial pressure and vital capacity after breast cancer surgery.

Design: Prospective cohort study participate in studies. Method: Blood gas measurements and Lung function (Vital capacity and FEV1) The day before surgery, the day after surgery and at follow-up.

Power analysis: There is a need to investigate 27 patients if the mean (SD) difference is 0.5 (1) kilopascal. Due to drop-outs the investigators calculate a need to include up to 60 patients.

ELIGIBILITY:
Inclusion Criteria:

• Women scheduled for surgery because of breast cancer.

Exclusion Criteria:

• Dementia or cognitive impairment that makes it impossible to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer scheduled for surgery.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen partial pressure | 1 day
  Change in oxygen partial pressure after surgery

SECONDARY OUTCOMES:
Carbon dioxide partial pressure | 1 day
  Change in carbon dioxide partial pressure after surgery
Vital capacity | 1 day
  Change in vital capacity after surgery
Forced expiratory volume in 1 second (FEV1) | 1 day
  Change in FEV1 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, MD, Prof, Principal Investigator — Dept Surgery, University hospital, Umea, Sweden
Locations (1):
- Dept of Surgery, University hospital, Umeå, Västerbotten County, Sweden